CLINICAL TRIAL: NCT00461487
Title: Reducing Teen Sexual Behavior: A Clinic-Based Approach
Brief Title: A Parent-Based Intervention to Reduce Sexual Risk Behavior in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AAAC1456; R34MH078719 (NIH); DAHBR 9A-ASAP
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: Adolescent Behavior; Communication; Health Behavior; Risk-Taking; Sexual Behavior
MeSH Terms: conditions — Behavior; Adolescent Behavior; Communication; Health Behavior; Risk-Taking; Sexual Behavior | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive sex education information during the physical exam
  Interventions: Behavioral: Families Talking Together
- 2 (Active Comparator): Participants will receive information on hygiene and nutrition during the physical exam
  Interventions: Behavioral: Active control on hygiene and nutrition
- 3 (No Intervention): Passive control participants will not receive any additional information during the physical exam

INTERVENTIONS:
Behavioral: Active control on hygiene and nutrition — The active control group will take place in a primary healthcare clinic and will be coordinated through allied health professionals when physicians see youth for their annual physical examination. The mother of the adolescent will meet with a social work interventionist for approximately 25 minutes while her child is being examined by the physician. During this time, the active control on hygiene and nutrition will be delivered to the mother.
  Arms: 2
Behavioral: Families Talking Together — The intervention will take place in a primary healthcare clinic and will be coordinated through allied health professionals when physicians see youth for their annual physical examination. A mother of the adolescent will meet with a social work interventionist for approximately 25 minutes while her child is being examined by the physician. During this time, the intervention will be delivered to the mother. At the conclusion of the session, the mother will be given reference materials to take home and tasks to perform to facilitate discussions about sex with her adolescent. There will be three follow-up booster sessions administered through phone calls to increase completion probabilities of the tasks. The target behavior is sexual activity in adolescents.
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of a parent-based intervention in reducing sexual risk behavior in high-risk Latino and African-American adolescents.

DETAILED DESCRIPTION:
In the United States, racial and ethnic minorities suffer disproportionately from preventable diseases and conditions. Many of these problems result from health-related behaviors that are established during childhood and adolescence. Latino and African-American adolescents are at considerable risk for the negative health consequences of early, risky sexual activity. This study will focus on inner-city Latino and African-American adolescents in grades 6, 7, and 8. The primary aim will be to develop an intervention that parents can use to address the issue of sexual risk behavior with their children.

The intervention will take place in a primary health care clinic when mothers accompany their children for annual physical exams. Mothers will meet with a social worker for approximately 25 minutes while their children are being examined by the physician. During this time, mothers will receive information about the problem of premature adolescent sexual activity, support in preventing or reducing their children's sexual risk behavior, instruction about how to talk with their children about sexual risk behavior, and targeted homework activities. All parents will also receive three follow-up phone calls to increase the probability that the homework tasks will be completed.

Participants in this study will also be assigned to one of the following three groups: an experimental group; an active control group; or a passive control group. Participants in all groups will complete three questionnaires over the course of the study to assess outcomes. Participants in the experimental and active control groups will partake in an additional meeting with a clinic social worker. Parents in the experimental group will meet with the social worker to discuss effective parent-adolescent communication strategies. They will also receive take-home materials to help them communicate with and parent their adolescents to reduce sexual risk behavior. Parents in the active control group will meet with the social worker to discuss adolescent nutrition and receive informational brochures.

Three booster sessions will take place via telephone for parents in the experimental and active control groups. The first booster call will occur approximately 1 month after study entry, the second will occur 5 months after the intervention ends, and the third will occur 9 months post intervention. No such booster calls will be provided to parents in the passive control condition.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent must be between the ages of 11 and 14 years old, and in grades 6, 7, or 8
* Adolescent is able to agree to being a participant
* Able to participate in questionnaire and intervention activities
* Latino or African-American descent

Exclusion Criteria:

* Any cognitive or psychiatric disability that would prevent successful participation in questionnaires and intervention activities

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 530 (Actual)
Dates: Start 2007-04; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Incidence of vaginal sexual intercourse measured | Measured at Months 3 and 12 post-treatment

SECONDARY OUTCOMES:
Incidence of condom use | Measured at Months 3 and 12 post-treatment
Incidence of oral sex | Measured at Months 3 and 12 post-treatment
Incidence of anal sex | Measured at Months 3 and 12 post-treatment
Number of sexual partners | Measured at Months 3 and 12 post-treatment
Behavioral intentions | Measured at Months 3 and 12 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Guilamo-Ramos, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University School of Social Work, New York, New York, United States

REFERENCES:
- [Derived] Guilamo-Ramos V, Bouris A, Jaccard J, Gonzalez B, McCoy W, Aranda D. A parent-based intervention to reduce sexual risk behavior in early adolescence: building alliances between physicians, social workers, and parents. J Adolesc Health. 2011 Feb;48(2):159-63. doi: 10.1016/j.jadohealth.2010.06.007. PMID 21257114